CLINICAL TRIAL: NCT06654687
Title: Transthoracic Echocardiographic Monitoring of Cardiac Output Effects of Colloid Preload and Crystalloid Coload During Cesarean Delivery Under Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sameh Fathy (Other)
Responsible Party: Sponsor-Investigator, Sameh Fathy, Assistant Professor of Anesthesia and ICU - Faculty of Medicine - Mansoura University, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ECHO for CO monitoring in CD
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Pregnancy; Cesarean Delivery; Spinal Anesthesia Induced Hypotension; Cardiac Output Measurement; Volume Status
Keywords: Cardiac output- Transthoracic ECHO - Colloids - Crystalloids - Cesarean delivery - Spinal anesthesia
MeSH Terms: interventions — Echocardiography; Ringer's Lactate; Albumins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crystalloid group (Active Comparator): Transthoracic Echocardiography will be used to measure the changes in stroke volume and cardiac output.
  Patients will receive 1000 mL of Ringer's lactate solution over 15 minutes.
  Interventions: Device: Transthoracic Echocardiography; Drug: Ringer lactate 1000 ml
- Combination group (Active Comparator): Transthoracic Echocardiography will be used to measure the changes in stroke volume and cardiac output.
  Patients will receive 250 mL of human albumin 5% over 10 minutes and 750 mL of Ringer's lactate solution over 15 minutes.
  Interventions: Device: Transthoracic Echocardiography; Drug: Albumin; Drug: Ringer lactate 750 ml

INTERVENTIONS:
Device: Transthoracic Echocardiography — Transthoracic Echocardiography will be used to measure the changes in stroke volume and cardiac output.
Drug: Ringer lactate 1000 ml — Patients will receive 1000 mL of Ringer's lactate solution over 15 minutes.
  Arms: Crystalloid group
Drug: Albumin — Patients will receive 250 mL of human albumin 5% over 10 minutes
  Arms: Combination group
Drug: Ringer lactate 750 ml — Patients will receive 750 mL of Ringer's lactate solution over 15 minutes.
  Arms: Combination group

SUMMARY:
Transthoracic echocardiography (TTE) has been introduced in anesthesia and intensive care practice to assess the volume status and predict fluid responsiveness, with a few studies performed on pregnant women (5).

In this study, we aim to evaluate the effect of intravenous administration of albumin as a colloid preload on the maternal stroke volume (SV) and cardiac output (CO) versus crystalloid coload. We used TTE to measure the changes in SV, and CO at baseline and at subsequent time points after spinal anesthesia.

DETAILED DESCRIPTION:
This prospective randomized controlled, double-blind study will be conducted at the obstetrics and gynecology operation room, at Qassim University Medical City.

Written informed consent will be obtained from eligible subjects on the day of the surgery. The study subjects will be randomized using the R software, version 3.5.2 (R Core Team, 2018; R Foundation for Statistical Computing, Vienna, Austria). Subjects will randomly be assigned to 2 equal groups (combined and crystalloid coload) using the permuted block randomization method with randomly selected block sizes of 4 and 6. The group allocation codes will be hidden in sequentially numbered, opaque, sealed envelopes that will be opened only after assessing the eligibility and obtaining the consent from the subjects. The study subjects and the outcome assessors will be blinded to the study group.

Spinal anesthesia will be conducted will be assessed respectively by an anesthesiologist not involved in the study.

All transthoracic cardiography images will be obtained by the second investigator who have the experience of accomplishing > 500 cases before starting the study using the technique and guidelines reported in American Society of Echocardiography . During obtaining the images intraoperatively, the investigator will be separated from the surgical field by a sterile drape, and the ultrasound probe will be covered with a sterile cover.

The study subjects will enter the operating room, lying supine on the operating table with slight left lateral position by tilting the operating table to the left. Standard monitors will be attached to all patients (noninvasive blood pressure, pulse oximeter, and electrocardiography). Basal systolic blood pressure and heart rate will be recorded after a period of rest, the average of 3 readings, 2 minutes apart will be recorded. Basal transthoracic cardiography images will be obtained.

Two 18-gauge intravenous cannula will be inserted in two large veins of the right forearm, one for IV fluids, and the other for phenylephrine infusion. In the combination group, patients will receive 250 mL of human albumin 5% (Human Albumin 50 gm/L, BAXTER, Austria) immediately before induction of spinal anesthesia (SA), over 10 minutes using an infusion pump (Fresenius Kabi Agilia Volumat MC Infusion Pump, Germany), and 750 mL of Ringer's lactate solution, to be started during the intrathecal injection of the local anesthetic, and infused over 15 minutes. In the crystalloid coload group, patients will receive 1000 mL of Ringer's lactate solution, to be started during the intrathecal injection of the local anesthetic, and infused over 15 minutes. In both groups, phenylephrine infusion will be given prophylactically, and will be started during the intrathecal injection of the local anesthetic at a dose ranging from 25-50 mcg/minute to maintain the SBP within 20 % of the basal readings. After administering the study solutions, Ringer's lactate will be attached to the IV cannula and will be administered at a rate of 1 mL/min; no other fluids will be administered until clamping of the umbilical cord (end of the study period).

In the sitting position, spinal anesthesia will be conducted by intrathecal injection of hyperbaric bupivacaine 12.5 mg 0.5% and fentanyl 15 microgram, using 27-gauge pencil point spinal needle at L3-L4 intervertebral space.

Surgery will be started after reaching at least an upper sensory level of T4; below this level, spinal anesthesia will be considered failed and patients will be excluded from the study.

SV and CO will be measured at 5 time points (basal readings, 1 minute after SA, 5 minutes after SA, immediately after delivery of the baby and clamping the cord, and 1 hour after the end of the study). SBP and HR will be recorded ever minute till the delivery of the baby, then every 3 minutes till the end of the surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status II parturients with full term singleton pregnancies scheduled for elective cesarean delivery under spinal anesthesia.

Exclusion Criteria:

* Height <150 cm, weight <55 kg, and body mass index ≥40 kg/m2.
* Women presenting in labor or having any contraindication to spinal anesthesia (patient refusal, increased intracranial pressure, coagulation disorders, or local skin infection).
* Chronic or pregnancy-induced hypertension; baseline systolic blood pressure >140 mm Hg.
* Hemoglobin <10 g/dL.
* Diabetes mellitus.
* Cardiovascular, cerebrovascular, or renal disease.
* Polyhydramnios or fetal abnormalities.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 162 (Actual)
Dates: Start 2024-10-27 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Changes in Cardiac Output | Immediately after delivery of baby
  The changes in Cardiac Output are measured relative to baseline immediately after delivery

SECONDARY OUTCOMES:
Changes in stroke volume | Immediately after delivery of baby
  The changes in stroke volume are measured compared to the baseline immediately after delivery
Total phenylephrine dose (mg) | Until delivery of baby
Total ephedrine dose (mg) | Until delivery of the baby
Total glycopyrrolate dose (mg) | Until delivery of the baby
Incidence of hypotension | Until end of surgery
  Decrease in SBP > 20% of the basal reading
Incidence of bradycardia | Until end of surgery
  Heart rate < 50 beats/minute
Incidence of nausea and/or vomiting | Until end of surgery
Measurement of APGAR score | 1 minute and 5 minutes after delivery of the baby
  APGAR score includes appearance, pulse, grimace, activity and respiration
Measurement of Urine output (ml) | 1 hour after delivery of the baby

CONTACTS AND LOCATIONS:
Overall Officials: MOHAMED TOLBA ELMORSY, MD, Principal Investigator — Lecturer of Anesthesia and ICU - Faculty of Medicine - Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Porter TR, Shillcutt SK, Adams MS, Desjardins G, Glas KE, Olson JJ, Troughton RW. Guidelines for the use of echocardiography as a monitor for therapeutic intervention in adults: a report from the American Society of Echocardiography. J Am Soc Echocardiogr. 2015 Jan;28(1):40-56. doi: 10.1016/j.echo.2014.09.009. No abstract available. PMID 25559474
- [Background] Rudski LG, Lai WW, Afilalo J, Hua L, Handschumacher MD, Chandrasekaran K, Solomon SD, Louie EK, Schiller NB. Guidelines for the echocardiographic assessment of the right heart in adults: a report from the American Society of Echocardiography endorsed by the European Association of Echocardiography, a registered branch of the European Society of Cardiology, and the Canadian Society of Echocardiography. J Am Soc Echocardiogr. 2010 Jul;23(7):685-713; quiz 786-8. doi: 10.1016/j.echo.2010.05.010. No abstract available. PMID 20620859
- [Background] McDonald S, Fernando R, Ashpole K, Columb M. Maternal cardiac output changes after crystalloid or colloid coload following spinal anesthesia for elective cesarean delivery: a randomized controlled trial. Anesth Analg. 2011 Oct;113(4):803-10. doi: 10.1213/ANE.0b013e31822c0f08. Epub 2011 Sep 2. PMID 21890886
- [Background] Practice Guidelines for Obstetric Anesthesia: An Updated Report by the American Society of Anesthesiologists Task Force on Obstetric Anesthesia and the Society for Obstetric Anesthesia and Perinatology. Anesthesiology. 2016 Feb;124(2):270-300. doi: 10.1097/ALN.0000000000000935. No abstract available. PMID 26580836
- [Background] Mercier FJ. Fluid loading for cesarean delivery under spinal anesthesia: have we studied all the options? Anesth Analg. 2011 Oct;113(4):677-80. doi: 10.1213/ANE.0b013e3182245af4. No abstract available. PMID 21948275
- [Background] Loubert C. Fluid and vasopressor management for Cesarean delivery under spinal anesthesia: continuing professional development. Can J Anaesth. 2012 Jun;59(6):604-19. doi: 10.1007/s12630-012-9705-9. Epub 2012 Apr 24. English, French. PMID 22528166